CLINICAL TRIAL: NCT00629265
Title: Efficacy of Electrical Stimulation for Dysphagia in Head & Neck Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: Northwestern University (Other); Boston University (Other); University of Wisconsin, Madison (Other); New York University (Other); VA Boston Healthcare System (U.S. Federal Agency); Lahey Clinic (Other); Lenox Hill Hospital (Other); Beth Israel Medical Center (Other); Greater Baltimore Medical Center (Other); Henry Ford Hospital (Other); University of California, San Diego (Other); University of Washington (Other); Mayo Clinic (Other); Icahn School of Medicine at Mount Sinai (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Susan Langmore, Director, Speech Language Pathology, Boston Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-26283; 5R01CA120950 (NIH)
Record Dates: First submitted 2008-01-30; First posted 2008-03-05 (Estimated); Results first posted 2014-10-31 (Estimated); Last update posted 2014-10-31 (Estimated); Status verified 2014-10

CONDITIONS: Dysphagia
Keywords: Dysphagia; Neuromuscular Electrical Stimulation (NMES); Head & Neck Cancer; Radiation and ChemoTherapy
MeSH Terms: conditions — Deglutition Disorders; Head and Neck Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active NMES + Swallowing Exercise (Active Comparator): Active Neurotech NT2000 Neuromuscular Electrical Stimulation (NMES) therapy will be paired concomitantly with repeated effortful sallowing exercises, for 60 swallows, 2 times per day, 6 days per week, for 12 weeks.
  Interventions: Device: Neurotech NT2000 Neuromuscular Electrical Stimulation (NMES)
- Sham NMES + Swallowing Exercise (Sham Comparator): Sham (inactive) Neurotech NT2000 Neuromuscular Electrical Stimulation (NMES) therapy will be paired concomitantly with repeated effortful sallowing exercises, for 60 swallows, 2 times per day, 6 days per week, for 12 weeks.
  Interventions: Device: Neurotech NT2000 Neuromuscular Electrical Stimulation (NMES)

INTERVENTIONS:
Device: Neurotech NT2000 Neuromuscular Electrical Stimulation (NMES) — NMES or Sham NMES will be paired with repeated, effortful swallowing behavior, for 60 swallows, 2 times a day, 6 days a week, for 12 weeks.
  Other Names: E-Stim; Neurotech NT2000

SUMMARY:
The purpose of the investigation is to learn whether intense swallowing exercise or intense swallowing exercise coupled with electrical stimulation (E-Stim) helps patients who had head/neck cancer and currently have dysphagia swallow better.

DETAILED DESCRIPTION:
Head and neck cancer patients have a better chance of survival in the 21st century because of radiation therapy (RT), either alone or in combination with surgery and/or chemotherapy (CRT). Such therapy has a high rate of local / regional control, and may extend duration of life. Unfortunately the elimination of the cancer can leave devastating side effects, including the inability to eat and swallow normally. Organ preservation, often assumed to be the preferred treatment, has now been shown to magnify dysphagia. Incidence of dysphagia in this group of patients is extremely high, with symptoms continuing to deteriorate for several years after treatment. Conventional therapy for dysphagia yields only minor benefit. Persistence of dysphagia has a major impact on the quality of life of these cancer survivors.

Recently, a new therapy approach has been introduced for dysphagia, called e-stim or Neuromuscular Electrical Stimulation (NMES). Through low voltage current delivered through the skin, motor nerves are excited, causing muscle contraction. An aggressive marketing campaign has turned e-stim into a very popular and sought-after therapy for dysphagia. However, there are no efficacy studies demonstrating its true benefit.

We have collected preliminary data with Head & Neck cancer patients using this modality and have seen improved swallow function in 9/15 patients. This is extremely promising and supports the need for a randomized clinical trial. The randomized controlled trial (RCT) proposed here will compare NMES therapy combined with exercise therapy to a sham NMES protocol combined with the same exercise therapy.

These therapies will be given to post-radiated H&N cancer patients who have moderate to severe dysphagia at least 3 months post-XRT (or post-XRT + post-CRT), to determine whether NMES is efficacious. Therapy will continue for 12 weeks with an intense, daily home program. Objective indicators of a change in swallow function will be taken from modified barium swallow (MBS) studies. Subjective measures of change will be the patients' self-reported diet, eating ability, and quality of life, and will indicate whether they perceived a benefit from the therapy.

This new treatment may represent the first real hope for improved swallowing in this growing population of cancer survivors. We need to determine whether it represents a truly beneficial treatment or whether our resources should be redirected. If successful, this study will stimulate a multitude of additional research to elucidate the mechanisms underlying this new treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ages 21+
* At least 3 months post-radiation therapy for head & neck cancer
* Treatment for their cancer can include chemotherapy.
* Surgery for their cancer, if done, must meet these criteria:

  * diagnostic biopsy
  * less than ½ of oral tongue resected
  * less than ½ of tongue base resected
  * no floor of mouth muscles resected
  * less than 50% of any other part of the oral cavity, pharynx or larynx resected
  * no resection of hyoid
  * Neck dissection, unilateral or bilateral neck dissections may have been completed prior to or after radiation therapy.
* Currently free of cancer, confirmed by head and neck exam within 2 months of beginning the study
* MBS demonstrates penetration or aspiration on at least one swallow during the study (minimum PAS = 4)
* The patient is free of any medical conditions that could limit the patient's ability to follow the protocol.
* No history of any swallowing problems prior to the onset of head and neck cancer
* Prior swallow therapy, if given to the patient, is neither an Inclusion nor Exclusion criteria

Exclusion Criteria:

* Inability to cooperate with the examination and treatment.
* An implanted electrical device (e.g., pacemaker, deep brain stimulator, defibrillator, vagal nerve stimulator)
* Previous e-stim treatment to the head & neck
* Any current or previous neurological disease which may adversely affect swallowing.
* History of oropharyngeal swallowing disorder prior to cancer.
* History of pre-cancer oral intake that was limited due to a swallowing problem.
* Previous neurosurgery on the brain that could compromise swallowing or ability to follow protocol.
* Severe COPD (oxygen dependent).
* Need for dilation of the upper esophageal sphincter or esophagus at time of entry.
* Females who are currently pregnant will be excluded from participation.
* Females of childbearing potential must have a negative pregnancy test and must be practicing a medically accepted means of contraception (including, but not limited to, condoms, diaphragms/caps, contraceptive pills, contraceptive rings/patches, intrauterine devices, hysterectomy or abstinence)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2008-03; Primary Completion 2012-04 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Langmore, PhD,SLP,BRS, Principal Investigator — Boston University
Locations (14):
- United States (14):
  - Mayo Clinic, Scottsdale, Arizona
  - University of California, San Diego, San Diego, California
  - Northwestern University, Evanston, Illinois
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Lahey Clinic, Burlington, Massachusetts
  - VA Boston Healthcare, West Roxbury, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Beth Israel Medical Center, New York, New York
  - New York University, New York, New York
  - Lenox Hill Hospital, New York, New York
  - Mout Sinai Medical Center, New York, New York
  - University of Washington, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 170 subjects were recruited/randomized into the study from 16 medical centers in the United States between January 2009 and December 2011. The majority of subjects were recruited during follow up visits in outpatient Otolaryngology & Radiation Oncology clinics.
Pre-assignment Details: All potentially eligible patients were screened with a 19 question eligibility form. 488 patients were screened, of which 318 were not eligible or declined to participate. 170 patients were then randomized to either the Active NMES + Swallowing Exercise group or the Sham (inactive) NMES + Swallowing Exercise group.
Groups:
- Active NMES + Swallowing Exercise: Active NMES paired concomitantly with repeated, effortful swallowing exercises, for 60 swallows, 2 times a day, 6 days a week, for 12 weeks.
- Sham NMES + Swallowing Exercise: Sham (inactive) NMES paired concomitantly with repeated, effortful swallowing exercises, for 60 swallows, 2 times a day, 6 days a week, for 12 weeks.
Period: Overall Study
Arm/Group | Active NMES + Swallowing Exercise | Sham NMES + Swallowing Exercise
Started | 116 | 54
Completed | 84 | 34
Not Completed | 32 | 20
Not completed — Lost to Follow-up | 4 | 5
Not completed — Withdrawal by Subject | 11 | 8
Not completed — Death | 1 | 0
Not completed — Adverse Event | 2 | 0
Not completed — HNC Recurrence | 4 | 0
Not completed — Other CA Requiring Treatment | 1 | 3
Not completed — Needed Esophageal Dilation | 4 | 1
Not completed — Unrelated Medical Complications | 3 | 1
Not completed — Unknown Reason | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Active NMES Group: NMES therapy combined with exercise therapy
- Sham NMES Group: Sham NMES combined with exercise therapy
- Total: Total of all reporting groups
Arm/Group | Active NMES Group | Sham NMES Group | Total
Number analyzed (Participants) | 116 | 54 | 170
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.1 (9.2) | 61.5 (10.6) | 61.9 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 9 | 25
  Male | 100 | 45 | 145
Region of Enrollment [Number; unit: participants]
  United States | 116 | 54 | 170

OUTCOME MEASURES:

1. Primary Outcome: Change in Penetration-Aspiration Scale (PAS) Score
Description: The PAS scale is a validated 8-point ordinal scale (Rosenbek et. al 1996) in which a score of 1 is best (material does not enter the airway) and a score of 8 is worst (material enters the airway, passes below the vocal folds, and no effort is made to eject it).
  Difference in mean PAS scores after 12 weeks of therapy was analyzed between the two groups of interest: Active NMES + Swallowing Exercise versus Sham (inactive) NMES + Swallowing Exercise. PAS scores were obtained from fluoroscopy (modified barium swallow) studies adminstered at three time points - enrollment, midway through treatment (6 weeks), and at end of treatment (12 weeks). All fluoroscopy studies were sent to, and analyzed by, a blinded external central laboratory.
Time Frame: Before and after treatment
Population: Note: the number of participants analyzed (125) does not match the total number enrolled (170) because 45 people did not have adequate follow up data required for this primary analysis.
Measure: Mean (Standard Deviation); unit: Change in points on PAS
Groups:
- Sham (Inactive) NMES + Swallowing Exercise: Sham (inactive) NMES paired concomitantly with repeated, effortful swallowing exercises, for 60 swallows, 2 times a day, 6 days a week, for 12 weeks.
Arm/Group | Active NMES + Swallowing Exercise | Sham (Inactive) NMES + Swallowing Exercise
Number analyzed (Participants) | 90 | 35
Change in points on PAS | 0.01 (1.04) | -0.57 (1.62)

2. Secondary Outcome: Performance Status Scale for Head and Neck Cancer Patients (PSS); The Head and Neck Cancer Inventory (HNCI)
Description: Perceive improved in quality of life and eating ability as measured by 2 validated scales: the Performance Status Scale for Head and Neck Cancer Patients (PSS) and The Head and Neck Cancer Inventory (HNCI).
  The PSS (List, et. al., 1990) is a clinician adminsitered scale that has three domains (normalcy of diet, eating in public, and understandability of speech). Each domain as well as overall score is scored on a scale of 0-100, with 0=worst and 100=best.
  The HNCI (Funk, et. al., 2003) is patient administered questionnaire that has four domains (social disruption, aesthetics, speech, eating). Each domain as well as overall score is scored on a scale of 0-100, with 0=worst and 100=best.
Time Frame: Before and after treatment
Population: Note: the number of participants analyzed (126) does not match the total number enrolled (170) because 44 people did not have adequate follow up data required for this secondary analysis.
Measure: Mean (Standard Deviation); unit: Change in PSS and HNCI score
Arm/Group | Active NMES + Swallowing Exercise | Sham (Inactive) NMES + Swallowing Exercise
Number analyzed (Participants) | 91 | 35
Change in PSS and HNCI score
  Change in Total PSS score | 6.25 (14.45) | 4.52 (16.06)
  Change in HNCI Eating Domain | 6.31 (17.92) | 6.74 (15.59)

ADVERSE EVENTS:
Time Frame: 3 years, 4 months
Arm/Group | Active NMES + Swallowing Exercise | Sham (Inactive) NMES + Swallowing Exercise
Serious Adverse Events (participants affected / at risk) | 14/116 | 5/54
Other Adverse Events (participants affected / at risk) | 12/116 | 7/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active NMES + Swallowing Exercise (N=116) | Sham (Inactive) NMES + Swallowing Exercise (N=54)
Death (General disorders) | 2 (2) | 0 (0)
Cancer Recurrence in Head & Neck (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0) — Two were base of tongue recurrances and one was a begnign vocal polyp
New Cancer / METs (other than Head & Neck) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Excision of Necrotic Mass (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Airway obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute allergic reaction to cat (Immune system disorders) | 0 (0) | 1 (1)
Lung biopsy for suspicious mass (Surgical and medical procedures) | 1 (1) | 0 (0)
PEG Complications (Gastrointestinal disorders) | 2 (2) | 0 (0) — 1 patient had an infection at PEG site and another had a blocked PEG
Blood pressure complications (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Dehydration requiring hospitilization (General disorders) | 1 (1) | 0 (0)
Exacerbation of COPD (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Progressive shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Laryngeal edema had been getting worse since end of RT and progressed to critical stage while in the study.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active NMES + Swallowing Exercise (N=116) | Sham (Inactive) NMES + Swallowing Exercise (N=54)
Tongue tingling / edema (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Severe Heartburn (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pain / discomfort in neck / throat (Musculoskeletal and connective tissue disorders) | 4 (5) | 1 (1)
Coughing (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Blood in sputum (General disorders) | 1 (1) | 0 (0)
Common Cold / Fever / Not Feeling Well (General disorders) | 2 (2) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bronchoscopy for RLL infiltrate (Surgical and medical procedures) | 1 (1) | 0 (0)
Patient over-medicated (General disorders) | 1 (1) | 0 (0)
Unable to tolerate electrode placement it c/o dizziness (General disorders) | 0 (0) | 1 (1)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Difficulty breathing d/t glottic stenosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pain related to oral biopsy (General disorders) | 1 (1) | 0 (0)
Lung biopsy for suspicious mass (Surgical and medical procedures) | 1 (1) | 0 (0)
Worstening of swallow - more difficult (Gastrointestinal disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Because of funding limitations research assistants could not be hired at most sites, and so 170 (instead of 240) subjects were enrolled. However, the results suggest additional patients would not have changed the outcome.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No